CLINICAL TRIAL: NCT03159000
Title: Double-Blind, Placebo Controlled Trial of Greater Occipital Nerve Block for the Treatment of Migraine Attacks
Brief Title: A Research Study of Greater Occipital Nerve Block as a Treatment for Acute Migraine Attacks
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Project never started - lack of resources and no subjects enrolled
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GON/WBY/003
Record Dates: First submitted 2017-04-26; First posted 2017-05-18 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Sodium Chloride; Lidocaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- GONB of lidocaine/bupivacaine (Experimental): The injectors will infiltrate an area of 2cm along the occipital ridge centering around the occipital artery or around the site 1/3 from the mastoid to the inion bilaterally. The subject will remain in the office for 30 minutes after injection, and receive a questionnaire to be filled out at 10 and 30 minutes, and 2 and 24 hours post-injection. Subjects who are not improved after 2 hours will be allowed to use their abortive treatment.
  Interventions: Combination Product: lidocaine/bupivacaine
- Placebo injection of 1/3 saline (Placebo Comparator): The injectors will infiltrate an area of 2cm along the occipital ridge centering around the occipital artery or around the site 1/3 from the mastoid to the inion bilaterally. The subject will remain in the office for 30 minutes after injection, and receive a questionnaire to be filled out at 10 and 30 minutes, and 2 and 24 hours post-injection. Subjects who are not improved after 2 hours will be allowed to use their abortive treatment.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Saline — 1ml of 1/3 saline
  Arms: Placebo injection of 1/3 saline
Combination Product: lidocaine/bupivacaine — 1ml of a 50% 2% lidocaine and 50% 0.5% bupivacaine
  Arms: GONB of lidocaine/bupivacaine

SUMMARY:
Several observational studies have shown improvement in episodic migraine with the use of greater occipital nerve block as an acute therapy, and a recent placebo controlled trial did not show a decrease in frequency of episodic or chronic migraine; however, there has never been a placebo controlled trial to investigate the efficacy of GONB as an acute treatment for headache, and there has been no determination of guidelines for selection of patients who would be most likely to respond to GONB. In light of the above, the investigators propose a double-blind, placebo-controlled, randomized trial examining the use of GONB with lidocaine/bupivocaine in patients with an acute episodic migraine. The results of this trial are expected to guide more appropriate therapeutic management of these participants and the optimal use of this procedure. 50 subjects will be entered into this study. This study is being conducted at Thomas Jefferson University only.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18 and 80 years old (inclusive) with a previous diagnosis fulfilling the international classification of headache disorders (ICHD3b) criteria for episodic migraine, presenting to clinic with an acute episodic migraine reported as at least a moderate pain level not lasting longer than 7 days at the time of injection.

Exclusion Criteria:

* subjects who have received greater occipital nerve block (GONB) in the past, subjects who in their own or the investigator's opinion are unable to describe their symptoms, subjects who have are scheduled to receive injection of onabotulinum toxin A within 72 hours, subjects who are pregnant or lactating.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects experiencing headache improvement at 2 hours | 2 hours
  Headache intensity on 4 point pain scale from moderate or severe to mild or none

SECONDARY OUTCOMES:
Percentage of subjects experiencing headache improvement 10 minutes | 10 minutes
  Headache intensity on 4 point pain scale from moderate or severe to mild or none.
Percentage of subjects experiencing headache improvement at 30 minutes | 30 minutes
  Headache intensity on 4 point pain scale from moderate or severe to mild or none.
Percentage of subjects experiencing headache improvement at 1 hour | 1 hour
  Headache intensity on 4 point pain scale from moderate or severe to mild or none.
Percentage of subjects experiencing headache improvement at 24 hours | 24 hours
  Headache intensity on 4 point pain scale from moderate or severe to mild or none.
Percentage of Subjects Achieving Resolution of Associated Symptoms of Nausea, Vomiting, Photophobia, Phonophobia, Osmophobia, Allodynia Measured at 10 minutes | 10 minutes
  Resolution of headache associated symptoms, including nausea, vomiting, photophobia, phonophobia, osmophobia and allodynia
Percentage of Subjects Achieving Resolution of Associated Symptoms of Nausea, Vomiting, Photophobia, Phonophobia, Osmophobia, Allodynia Measured at 30 minutes | 30 minutes
  Resolution of headache associated symptoms, including nausea, vomiting, photophobia, phonophobia, osmophobia and allodynia
Percentage of Subjects Achieving Resolution of Associated Symptoms of Nausea, Vomiting, Photophobia, Phonophobia, Osmophobia, Allodynia Measured at 1 hour | 1 hour
  Resolution of headache associated symptoms, including nausea, vomiting, photophobia, phonophobia, osmophobia and allodynia
Percentage of Subjects Achieving Resolution of Associated Symptoms of Nausea, Vomiting, Photophobia, Phonophobia, Osmophobia, Allodynia Measured at 2 hours | 2 hours
  Resolution of headache associated symptoms, including nausea, vomiting, photophobia, phonophobia, osmophobia and allodynia
Percentage of Subjects Achieving Resolution of Associated Symptoms of Nausea, Vomiting, Photophobia, Phonophobia, Osmophobia, Allodynia Measured at 24 hours | 24 hours
  Resolution of headache associated symptoms, including nausea, vomiting, photophobia, phonophobia, osmophobia and allodynia

CONTACTS AND LOCATIONS:
Overall Officials: William B Young, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No